CLINICAL TRIAL: NCT01693133
Title: A Multicenter, Prospective, Randomized, Controlled, Comparative Parallel Study of Dehydrated Human Amnion/Chorion Membrane (dHACM) Wound Graft in the Management of Diabetic Foot Ulcers
Brief Title: Trial of Dehydrated Human Amnion/Chorion Membrane (dHACM) In the Management of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFDFU003
Record Dates: First submitted 2012-09-19; First posted 2012-09-26 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Other): Standard of Care: Moist Wound Therapy and Offloading
  Interventions: Other: Standard of Care: Moist Wound Therapy and Offloading
- EpiFix plus Standard of Care (Experimental): Weekly application of EpiFix (up to 12 week) and standard of care (moist wound therapy and offloading)
  Interventions: Other: EpiFix plus Standard of Care

INTERVENTIONS:
Other: Standard of Care: Moist Wound Therapy and Offloading — Standard of Care: Moist Wound Therapy and Offloading
  Arms: Control
Other: EpiFix plus Standard of Care — Weekly application of EpiFix and Standard of Care
  Arms: EpiFix plus Standard of Care

SUMMARY:
The objective of this study is to evaluate the percentage of patients with complete diabetic foot ulcer (DFU) closure following up to 12 weeks of treatment with either dehydrated human amnion/chorion membrane (dHACM) plus standard of care (SOC) or SOC alone.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18 or older.
2. The patient is willing and able to provide informed consent and participate in all procedures and follow up evaluations necessary to complete the study.
3. Patient's ulcer must be diabetic in origin with a size ranging from 1 to 25 cm2. Debridement will be done prior to randomization, if clinically indicated.
4. Wounds should be diabetic foot ulcers located on the dorsal or plantar surface of the foot.
5. Patients with Type 1 or 2 diabetes (criteria for the diagnosis of diabetes mellitus per ADA).
6. Ulcer must be present for a minimum of 30 days before enrollment/randomization, with documented failure of prior treatment to heal the wound (≤25% wound area reduction after 14 consecutive days of therapy immediately prior to randomization when treated with standard protocol of care).
7. Affected leg has been offloaded (removable walker or total contact cast) for >14 consecutive days prior to randomization.
8. Serum Creatinine less than 3.0mg/dl (within last 6 months).
9. HbA1c less than 12% within previous 60 days.
10. Patient has adequate circulation to the affected extremity, as demonstrated by one of the following within the past 60 days:

    * Dorsum transcutaneous oxygen test (TcPO2) with results ≥30mmHg, OR
    * ABIs with results of ≥0.7 and ≤1.2, OR
    * Doppler arterial waveforms, which are triphasic or biphasic at the ankle of affected foot.
11. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence).

Exclusion Criteria:

1. Patients presenting with an ulcer probing to bone (UT Grade IIIA-D). A positive probe-tobone will be confirmed when bone or joint can be felt with a sterile, ophthalmological probe.
2. Patients with multiple wounds on the same foot where other wounds are within 3 cm of the wound under care.
3. Patients considered not in reasonable metabolic control, confirmed by an HbA1c 12% or greater at any time within previous 60 days.
4. Known history of poor compliance with medical treatments.
5. Patients currently enrolled in this study. Concurrent enrollment in the study is prohibited.
6. Patients treated with investigational drug(s) or therapeutic device(s) within 30 days.
7. Patients currently receiving radiation therapy or chemotherapy.
8. Known or suspected local skin malignancy to the index diabetic ulcer.
9. Patients diagnosed with autoimmune connective tissue diseases.
10. Non-revascularizable surgical sites.
11. Active infection at index site or currently being treated with antibiotics
12. Any pathology that would limit the blood supply and compromise healing.
13. Patients that have received a biomedical or topical growth factor for their wound within the previous 30 days. Study ulcer has been previously treated with tissue engineered materials (e.g. Apligraf® or Dermagraft®) or other scaffold materials (e.g. Oasis, Matristem) within the last 30 days.
14. Patients who are known to be pregnant, plan to become pregnant, or are breast feeding.
15. Known allergy to Gentamicin sulfate or Streptomycin sulfate.
16. Active Charcot deformity or major structural abnormalities of the foot.
17. Wounds that are greater than one year in duration without intermittent closure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2012-07; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with complete closure of the study ulcer | Week 12
  Assessed by the Investigator, during treatment (Visits 1 - 13).

SECONDARY OUTCOMES:
Time to complete closure for both groups | Up to 12 Weeks
  As assessed by photographic evaluation and the Investigator
Rate of wound closure | Up to Week 12
  As assessed by photographic evaluation and the Investigator
Incidence of ulcer recurrence | Up to Week 16
  Incidence of ulcer recurrence at the site of the study ulcer during the follow up phase.
Quality of Life | Up to Week 12
  Change in quality of life metrics as measured by SF-36 Health Survey and changes in the patient's reported pain scores as measured by the Visual Analog Scale.
Cost effectiveness of treatment | Up to Week 12
  Cost effectiveness of treatment regimen.

OTHER OUTCOMES:
Safety | Up to Week 16
  The Safety population will be used for the analysis of safety endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: William Tettelbach, MD, Principal Investigator — Intermountain Medical Center
Locations (20):
- United States (20):
  - Central Research Associates, Inc., Birmingham, Alabama
  - Stockdale Podiatry Group, Bakersfield, California
  - Center for Clinical Research Inc, Castro Valley, California
  - Valley Vascular Surgery Associates, Fresno, California
  - Limb Preservation Platform, Fresno, California
  - Novak Urgent Care and Family Practice, Indio, California
  - Loma Linda VA Medical Center, Loma Linda, California
  - Foot & Ankle Clinic, Los Angeles, California
  - Palmtree Clinical Research, Inc., Palm Springs, California
  - Center for Clinical Research, Inc., Sacramento, California
  - Center for Clinical Research, San Francisco, California
  - MetroWest Medical Center, Framingham, Massachusetts
  - South Shore Hospital, Weymouth, Massachusetts
  - Jobst Vascular Institute, Promedica Toledo Hospital, Toledo, Ohio
  - Center for Clinical Research, Inc., Eugene, Oregon
  - Dorn VA, Columbia, South Carolina
  - Futuro Clinical Trials, LLC, McAllen, Texas
  - IMC Wound Care, Murray, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Coastal Podiatry, Inc., Virginia Beach, Virginia